CLINICAL TRIAL: NCT03340753
Title: An Open-Label, Partial Crossover, Single-Dose Study to Evaluate the Pharmacokinetics, Dose-Proportionality, and Safety/Tolerability of Tablet Versus Capsule Formulations of KBP 5074 in Healthy Subjects
Brief Title: Bioavailability of KBP-5074 Tablet vs Capsule Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KBP5074-1-004
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bioequivalence
MeSH Terms: interventions — KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KBP-5074 Capsule (Active Comparator): KBP-5074 capsule, 0.5 mg or 1.0 mg, QD, single dose
  Interventions: Drug: KBP-5074 Capsule
- KBP-5074 Tablet (Experimental): KBP-5074 tablet, 0.5 mg or 1.0 mg, QD, single dose
  Interventions: Drug: KBP-5074 Tablet

INTERVENTIONS:
Drug: KBP-5074 Capsule — KBP-5074 (0.5 mg or 1.0 mg) capsule formulation single dose, in a 2-period crossover design with a 2-week washout/follow-up period
  Other Names: MRA
  Arms: KBP-5074 Capsule
Drug: KBP-5074 Tablet — KBP-5074 (0.5 mg or 1.0 mg) tablet formulation single dose, in a 2-period crossover design with a 2-week washout/follow-up period
  Other Names: MRA
  Arms: KBP-5074 Tablet

SUMMARY:
This is an open-label, partial crossover, single-dose study to evaluate the pharmacokinetics (PK), dose proportionality, and safety/tolerability of tablet versus capsule formulations of KBP-5074 in healthy subjects. The study is designed to evaluate the PK of a new tablet formulation versus that of the current capsule formulation. Data derived from this study, in addition to preclinical data and chemistry, manufacturing, and controls, will provide a basis for dose selection in future studies.

DETAILED DESCRIPTION:
Twenty healthy subjects will be allocated 4:1 to either the crossover study groups (16 subjects) or to the 0.25 mg tablet single dose treatment (4 subjects). Subjects allocated to the crossover study groups will be randomized 1:1 to 0.5 mg tablet/capsule (8 subjects) or 1.0 mg tablet/capsule (8 subjects).

Within the crossover study groups, subjects will be further randomized to receive a single dose of KBP-5074 (0.5 mg or 1.0 mg) in either capsule or tablet formulation in a 2-period crossover design with a 2-week washout period. The study duration for subjects in the crossover study groups will be approximately 7 weeks, which includes a 3-week screening period, and the 2 crossover single dose periods, which will be followed by a 2-week washout/follow-up period, respectively.

Subjects allocated to the 0.25 mg dose cohort (n=4) will receive a single dose of 0.25 mg in tablet formulation only. The 0.25 mg tablet cohort will provide additional data for the evaluation of dose exposure for the tablet formulation. The study duration for the single dose arm will be 5 weeks, which includes a 3-week screening period, and the single dose which will be followed by a 2 week washout period.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy male and females, aged 18 to 45, inclusive;
* Body mass index (BMI) between 18 to 30 kg/m2, inclusive;
* Nicotine-free (cigarettes, pipe, cigar, chewing tobacco, nicotine patches, etc.) for at least 6 months prior to Screening until the end of the study;
* Normal renal function as defined by estimated glomerular filtration rate >90 mL/min/1.73m2;
* Willing to remain in the study facility for the duration of the domicile period and able to return for all out-patient visits;
* Ability to understand and sign written informed consent, which must be obtained prior to any study-related procedures being completed;
* Willing to avoid adding salt substitutes that contain potassium chloride or potassium lactate to food from 7 days prior to dosing through the duration of the study;
* Women of childbearing potential (WOCBP), must agree to 2 medically accepted, effective methods of birth control during the study and for 90 days after the end of the study. Adequate methods of contraception are defined as those that result in a low failure rate (<1% per year) when used consistently and correctly. Such methods include the use of oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products (such as an intrauterine diaphragm, condoms, or spermicides);
* Women of childbearing potential are defined as women who are not surgically or chemically sterilized, including hysterectomy or bilateral oophorectomy (tubal ligation is not acceptable), and who are between menarche and 1 year post-menopause; and
* Post-menopausal is defined as amenorrhoeic for at least 1 year prior to screening AND, if aged under 45 years have a serum follicle stimulating hormone (FSH) level of at least 30 IU/L. Women who are taking hormone replacement therapy (HRT) do not have to have FSH assessments, but the amenorrhea (before starting HRT) must have been naturally (spontaneously) occurring and have been accompanied by an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms);
* Males with partners who are WOCBP must agree to use condoms plus spermicide and their female partner must also be using contraception (e.g., hormonal or intra-uterine device). This double contraception must be used from the first dose of study drug until at least 90 days after the last dose of study drug;
* Males must also refrain from donating sperm during the study and for 90 days after the last dose;
* Negative urine test for drugs of abuse (opiates, benzodiazepines, amphetamines, cannabinoids including tetrahydrocannabinol, cocaine, barbiturates, and phencyclidine), nicotine/cotinine, and breath alcohol test at Screening and Check-in; and
* Is in good general health as determined by the Investigator's review of medical history, concomitant medications, physical examination, and clinical laboratory and electrocardiogram (ECG) evaluations at the Screening Visit.

Exclusion Criteria:

* History of any illness, that, in the opinion of the Investigator, could confound the results of the study or pose an additional risk to the subject by their participation in the study ;
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease;
* Any surgical or medical condition that could interfere with the absorption, distribution, metabolism, or excretion of the IMP;
* History of any clinically significant drug allergy as per the Investigator's judgment;
* History of alcohol abuse or illicit drug use within 2 years of Screening;
* Use of marijuana (including prescribed marijuana) within 3 months prior to Screening;
* Use of nicotine within 6 months prior to screening;
* Use of any prescription or over-the-counter medication, vitamins/herbal supplements (with the exception of hormonal contraceptives or HRT and sporadic use of acetaminophen or ibuprofen) within 7 days (14 days if the drug is a potential enzyme inducer) prior to study allocation;
* Has taken any investigational medicinal product (IMP) within 30 days or 5 half-lives of that IMP (whichever is longer) prior to dosing;
* Donation of blood or blood products within 30 days of dosing;
* Acute illness within 14 days of dosing; acute illness occurring prior to the 14 days before dosing must show signs of complete recovery;
* Regular caffeine consumption of >300 mg/day (i.e., approximately 3 cups [8 fluid ounces] of coffee or 10 cans [12 fluid ounces] of cola) 7 days prior to dosing. Inability to restrict consumption of caffeine during the domicile period;
* Positive serologic findings for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV);
* Diets that could alter metabolism (i.e., vegetarian, high protein, Slim Fast®, Nutrisystem®, etc.) 7 days prior to dosing;
* Weight loss or gain of ≥10% in the 30 days prior to dosing;
* Strenuous exercise (>5 per week) within 2 weeks prior to dosing;
* Positive urinary cotinine level, breath alcohol, or drug screen at Screening and/or admission (both admissions for subjects in the crossover treatment group);
* Systolic BP >140 mmHg or <90 mmHg or diastolic BP >90 mmHg or <60 mmHg at Screening with 1 repeat allowed per Investigator discretion at Screening and Day -1 (and Day 14 for subjects in the crossover treatment group period 2);
* Heart rate <40 bpm or >100 bpm at Screening;
* Consumption of any nutrients known to modulate cytochrome P450 3A4 (CYP3A4) or any strong inhibitors or inducers of CYP3A4, starting from 14 days prior to the first dose of study drug at Day 1 until the end of study assessments. Inability to refrain from consumption of grapefruit and Seville oranges or St. John's wort (14 days prior to dosing and during the study);
* Positive pregnancy test result;
* Subject has any finding that, in the view of the Investigator and/or Medical Monitor, would compromise the subject's safety; or
* The Investigator has any reason to believe that the subject may be unable to fulfill the protocol visit schedule or requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
AUClast | Through 312 hours
  Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last quantifiable plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace CLinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No